CLINICAL TRIAL: NCT04227080
Title: To Evaluate BH4 Responsiveness in PAH Deficiency PKU Patients Who Failed to Achieve 30% Blood Phe Reduction Within 24-hour BH4 Loading Test by Extending the Period of BH4 Response Test: A Pilot Study in Taiwan
Brief Title: BH4 Responsiveness in PAH Deficiency PKU Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, vghtpe user, Chairman, Department of Pediatrics, Taipei Veterans General Hospital, Taiwan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0, 2018/03/21
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Pku Phenylketonuria; PAH Deficiency
Keywords: Phenylketonuria, PAH Deficiency, Kuvan
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: BH4 — oral administration of 20 mg/kg KUVAN (BH4)

SUMMARY:
Most forms of Phenylketonuria and hyperphenylalanemia are caused by mutations in the PAH gene (phenylalanine hydroxylase) which is responsible for the conversion of Phe into tyrosine, in the presence of the molecular oxygen and cofactor tetrahydrobiopterin (BH4). To prevent mental retardation due to the buildup of neurotoxic metabolites of Phe, patients with severe PKU must be treated with a low-Phe diet starting early in their life [1]. Although Phe-restricted diet control is essential for avoiding neurological impairment, the life-long compliance with this dietary control is not optimally maintained, particularly in adulthood and adolescence [2]. Non-adherence to dietary control after successful treatment in early childhood may contribute to lower intelligence quotient (IQ), emotional and behavioral disorders, including attention deﬁcit disorders, depression, anxiety, and agoraphobia.

In recent years, another therapeutic approach for managing PKU is to supplement a synthetic form of BH4 along with diet control. Kure et al. and several other research teams had indicated that treatment with BH4 might lower down the Phe level in a subset of PKU patients [3-7]. BH4 acts as a pharmacological chaperone to stabilize mutant enzymes with disrupted tetramer assembly and increased sensitivity to proteolytic cleavage and aggregation. The BH4-supplementation therapy (Kuvan) can be used to loosen or even replace burdensome dietary treatment of PKU patients. Correct and efficient identification of BH4-responsive patients is important, both to improve the fast assessment, as well as to avoid false expectations and unnecessary costs. Unfortunately, there is still no golden standard on how to assess BH4 responsiveness most efficiently.

In Taiwan, high-dose BH4 [20mg/kg] loading is the standard test to identify patients who are responsible to BH4 treatment, for PAH deficiency PKU patients with more than 30% decrease in Phe level within 24 hours after BH4 challenge were BH4-responsive patients and eligible for national health insurance coverage of continuous BH4 treatment. In clinical studies, blood Phe levels in patients who are BH4-responsive typically decrease within 24 hours after a single administration of Kuvan, although the maximal effect on blood Phe levels may take up to a month. A Phase IV open-label trial showed that of 64% of patients responded to Kuvan within 7 days whereas 10% responded between 8-28 days. To the best of our knowledge, there's no previous study which evaluated longer than 7 days BH4 response test in Asian countries, and for the purpose to help PAH deficiency PKU patients achieve optimal Phe control and neurocognitive outcomes, it's definitely worthy to extend the period of BH4 response test to identity more patients who can benefit from Kuvan treatment.

DETAILED DESCRIPTION:
Objectives

1. Changes of blood Phe level from baseline at the 7th, 14th, and 28th day
2. Percentage of the study patients whose blood Phe level decreases for >= 30%
3. Percentage of the study patients whose Phe tolerance increase from baseline for >=50%
4. Correlation between PAH gene mutation and blood Phe level reduction

Study Design and Methodology The PAH deficiency PKU patients who failed to achieve 30% blood Phe reduction within 24-hour BH4 loading test will be enrolled to this study. Baseline protein intake will be calculated and baseline blood phenylalanine levels will be established prior to starting the trial. During the entire testing period, patients will have no dietary restrictions. Blood Phe will be measured on day 1, 7, 14 and 28 days after oral administration of 20 mg/kg KUVAN in 40 patients whose initial plasma Phe results were ≥360 umol/L. In this study, the efficacy of BH4 will be evaluated on 7, 14 and 28 days to determine whether a patient is BH4-responsive. The total duration of patient participation in the study will be up to 3 months (1 month of BH4 efficacy evaluation and up to 8 weeks of screening).

* Health status assessments：A complete physical examination will be performed at all study visits. The physical examination will include appearance, eyes, ears, nose, head, throat, neck, chest, lungs, heart, abdomen, extremities, skin and musculoskeletal system. Weight will be measured at first visit, without shoes and having removed all outwear such as jackets, sweaters or sweatshirts and heavy pocket items. Clinically significant findings at screening will be reported as medical history and as adverse event after the screening visit.
* Vital sign：Vital signs measurement will be recorded at all study visits and will include body temperature, respiration, blood pressure and heart rate after the patients has sat quietly for at least 5 minutes.
* Nutrition assessment：Baseline protein intake will be calculated from 3-day photographic food records, and baseline blood Phe level will be established after a 3-5 hour fasting prior to starting BH4 loading. During the entire testing period, patients will have no dietary restrictions, but will be asked to keep a stable diet throughout the study. Patients will be required to keep a diary and photographic food records for three days of each week containing a record of all foods and beverages ingested including synthetic and low protein containing foods. Dietary records will be reviewed by a single qualified metabolic dietician and monitored for calorie intake, natural protein intake, synthetic protein intake, and total Phe intake.
* Laboratory assessments：All routine clinical laboratory assessments will be performed by central laboratory. The laboratory evaluations will include :

  * Serum nutritional biomarkers : total protein, albumin, total cholesterol, total triglyceride, LDL (low-density lipoprotein cholesterol), HDL (high-density lipoprotein cholesterol), Iron, Ferritin
  * Blood phenylalanine and tyrosine : Blood phenylalanine and tyrosine levels will be measured prior to BH4 loading test, and on day 1, 7, 14 and 28 days following kuvan 20 mg/kg/day.
  * PAH gene evaluation in all patients
  * Urine pTerin and DHPR enzyme activity analysis - Patients with defect in the synthesis and recycling of BH4 will be excluded by analysis of urinary pterins and dihydropteridine reductase activity in erythrocytes. pTerins (neopterin and biopterin) metabolism will be analyzed in each visit.
* Dispense study drug - Subjects will receive 20 mg/kg Kuvan administered orally once daily for 28 days.

ELIGIBILITY:
Inclusion criteria

1. Subjects have a confirmed diagnosis of PAH deficiency PKU, defined as baseline blood Phe levels of >360 umol/L
2. Subject and/or parent or guardian must be capable of understanding and providing written informed consent
3. For PAH deficiency PKU newborns, they should be identified as non-BH4 responders by 24-hour BH4 loading test after birth
4. For PAH deficiency PKU older pediatric and adult patients, they should be identified as non-BH4 responders by 24-hour BH4 loading test and currently use Phe-restricted diet control alone

Exclusion criteria

1. Perceived to be unreliable or unavailable for study participation or, if under the age of 18, had parents or legal guardians who the investigator perceived to be unreliable or unavailable
2. Used any investigational agent other than Kuvan within 30 days of screening, or required any investigational agent or investigational vaccine prior to completion of all scheduled study assessments
3. Pregnant or breastfeeding, or considering pregnancy
4. Concurrent disease or condition that would interfere with study participation or safety (eg, seizure disorder, asthma or other condition requiring oral or parenteral corticosteroid administration, insulin-dependent diabetes, or organ transplantation recipient)
5. Serious neuropsychiatric illness (eg, major depression) not currently under medical management
6. Required concomitant treatment with any drug known to inhibit folate synthesis (eg, methotrexate)
7. Clinical diagnosis of primary BH4 deficiency
8. Patients him/herself or his/her caregivers are unable or unwilling to sign informed consent or to comply with the requirements of the study
9. Patient attend other clinical trials should not be included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Changes of blood Phe level from baseline | 7th, 14th, and 28th day
  Changes of blood Phe level from baseline at the 7th, 14th, and 28th day

SECONDARY OUTCOMES:
Phe level decreases for >= 30% | 7th, 14th, and 28th day
  Percentage of the study patients whose blood Phe level decreases for >= 30%
Phe tolerance increase from baseline for >=50% | 7th, 14th, and 28th day
  Percentage of the study patients whose Phe tolerance increase from baseline for >=50%
PAH gene mutation and Phe level | 7th, 14th, and 28th day
  Correlation between PAH gene mutation and blood Phe level reduction